CLINICAL TRIAL: NCT01380587
Title: Utility of XCL1 as a Prognostic Marker in Acute Lymphoblastic Leukemia
Acronym: XCL1
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, MD, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: XCL1 in ALL
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; XCL1; Cytokines; Prognosis
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, blasts
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Lymphoblastic Leukemia: We will invite patients with newly diagnosed acute lymphoblastic leukemia in the Department of Hematology, who had not received anticancer therapy and regardless the subtype and immunophenotype of the disease.

SUMMARY:
The purpose of the study is to determine the utility of XCL1 in the prognosis of acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Each year approximately 256,000 children and adults around the world develop a form of leukemia, and 209,000 died from it. Recently, some studies have evaluated the relationship between the concentration of some cytokines and prognosis of acute lymphoblastic leukemia. XCL1 is a lymphotactin that belongs to a cytokine subfamily called C or γ with only one cysteine in the N-terminal residue. It has been found with significant expression of receptor mRNA XCL1 (XCR1) in T and B lymphocytes and related to hematological neoplasms. For these reasons, XCL1 could be a efficient marker of prognosis in patients with acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly diagnosed acute lymphoblastic leukemia .

Exclusion Criteria:

* Patients with prior treatment with chemotherapeutic agents.
* Patients treated with immunosuppressants.
* Patients under 12 months old.
* Patients with a diagnosis or history of autoimmune diseases.
* Patients with a diagnosis or history of immunosuppressive diseases.
* Patients who do not agree to sign a Letter of Informed Consent.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will invite patients with newly diagnosed acute lymphoblastic leukemia , who had not received anticancer therapy and regardless the subtype and immunophenotype of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with poor prognosis and high levels of XCL1 | 3 months
  Number of patients with high levels of XCL1, expression of its receptor and other cytokines.
Number of patients with poor prognosis and high levels of cytokines | 3 months
  Measurements obtained will be evaluated to assess the prognosis of patients and made correlations with the concentration of IL-1β, IL-2 and XCL1 as well as the relationship XCR1 XCL1 and in leukemic cells.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar H Gutierrez Aguirre, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez UANL
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Huang H, Li F, Cairns CM, Gordon JR, Xiang J. Neutrophils and B cells express XCR1 receptor and chemotactically respond to lymphotactin. Biochem Biophys Res Commun. 2001 Feb 23;281(2):378-82. doi: 10.1006/bbrc.2001.4363. PMID 11181058
- [Background] Taub DD, Oppenheim JJ. Chemokines, inflammation and the immune system. Ther Immunol. 1994 Aug;1(4):229-46. PMID 7584498
- [Background] Oppenheim JJ, Zachariae CO, Mukaida N, Matsushima K. Properties of the novel proinflammatory supergene "intercrine" cytokine family. Annu Rev Immunol. 1991;9:617-48. doi: 10.1146/annurev.iy.09.040191.003153. PMID 1910690
- [Background] Bazan JF, Bacon KB, Hardiman G, Wang W, Soo K, Rossi D, Greaves DR, Zlotnik A, Schall TJ. A new class of membrane-bound chemokine with a CX3C motif. Nature. 1997 Feb 13;385(6617):640-4. doi: 10.1038/385640a0. PMID 9024663
- [Background] Rollins BJ. Chemokines. Blood. 1997 Aug 1;90(3):909-28. No abstract available. PMID 9242519
- [Background] Stievano L, Tosello V, Marcato N, Rosato A, Sebelin A, Chieco-Bianchi L, Amadori A. CD8+ alpha beta+ T cells that lack surface CD5 antigen expression are a major lymphotactin (XCL1) source in peripheral blood lymphocytes. J Immunol. 2003 Nov 1;171(9):4528-38. doi: 10.4049/jimmunol.171.9.4528. PMID 14568926